CLINICAL TRIAL: NCT05906082
Title: Text-messaging E-cigarette Cessation Intervention for Young Adults in Rural Areas: A Pilot Study
Brief Title: Vape-Free Text-Messaging: Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jovan Gwon, PhD, RN, FIAAN (Other)
Responsible Party: Sponsor-Investigator, Jovan Gwon, PhD, RN, FIAAN, Associate Professor, University of Wisconsin, Milwaukee
Organization: University of Wisconsin, Milwaukee (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23.179
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: E-cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (E-cigarette cessation text-messaging intervention) (Experimental)
  Interventions: Behavioral: E-cigarette cessation text-messaging intervention
- Standard care (Standard care control using standard national resources) (Active Comparator): This standard care group will receive standard care resources from smokefree.gov.
  Interventions: Behavioral: Standard care control using standard national resources

INTERVENTIONS:
Behavioral: E-cigarette cessation text-messaging intervention — This is the intervention for e-cigarette cessation using text messages targeting young adults in rural areas.
  Arms: Intervention (E-cigarette cessation text-messaging intervention)
Behavioral: Standard care control using standard national resources — This is the standard care with national resources from smokefree.gov.
  Arms: Standard care (Standard care control using standard national resources)

SUMMARY:
This is a small pilot randomized controlled trial to evaluate the feasibility, acceptability, and preliminary efficacy of the e-cigarette cessation text-messaging intervention with young adults in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 18-24 years
* everyday e-cigarette use in the past month
* ownership of a mobile phone or smartphone with texting and internet access abilities
* knowledge of how to use text messages
* plan on quitting e-cigarette use within one month
* home address in a rural county of Wisconsin, Minnesota, North Dakota, and South Dakota

Exclusion Criteria:

* Individuals who reported use of other tobacco products (e.g., cigarettes, smokeless tobacco) than e-cigarettes in the past month

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited and randomized | Throughout 12 months
  Number of participants recruited and randomized
Self-reported proportion of text messages read | At 1 month
  Proportion of text messages read during the intervention or standard care at 1 month
Retention rates (proportion of participants remained until 1 month post-intervention from enrollment) | At 1 month
  Proportion of participants from enrollment to 1 month post-intervention or standard-care
Level of acceptability of the intervention | At 1 month
  1. When you had received our text messages from our VapeFreeTXT program 1 month ago, how many of our text messages did you read on a typical day? Not at all (1) Read about 25% messages (2) Read about half messages (3) Read about 75% messages (4) Read the entire messages (5)
  2. How useful was our VapeFreeTXT program in helping you quit vaping? Not at all useful (1) Slightly useful (2) Moderately useful (3) Very useful (4) Extremely useful (5)
  3. Did our VapeFreeTXT program make you think about quitting vaping? Not at all (1) Probably not (2) Neither yes nor no (3) Probably yes (4) Definitely yes (5)
  4. Do you think our VapeFreeTXT program will change your vaping? Not at all (1) Probably not (2) Neither yes nor no (3) Probably yes (4) Definitely yes (5)
  5. Would you recommend this program to a friend or others? Not at all (1) Probably not (2) Neither yes nor no (3) Probably yes (4) Definitely yes (5)
Proportion of salivary cotinine samples returned | At 1 month
  Proportion of salivary cotinine samples returned to the office lab for cotinine analysis
Self-reported 7-days point prevalence abstinence from ENDS and other tobacco | At 1 month
  Self-reported 7-days point prevalence abstinence from ENDS and other tobacco
Concentration of cotinine in saliva | At 1 month
  Biochemically verified abstinence evaluated by salivary cotinine samples
Nicotine dependence (Penn State Electronic Cigarette Dependence Index) | At 1 month
  Nicotine dependence (minimum 0 to maximum 20, higher scores mean a worse outcome.)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No